CLINICAL TRIAL: NCT03502720
Title: Analysis of a Customized Percutaneous External Guidance System for Scaphoid Fracture Fixation Using 3D Printing
Brief Title: A Personalised Percutaneous External 3D Guide for Scaphoid Fixation
Acronym: Scaphix
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Francesc A. Marcano-Fernández, MD, Corporacion Parc Tauli
Other Study IDs: CSPTCOT2018533
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Scaphoid Bone Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Patients: Data obtained retrospectively from Scaphoid fixation surgeries performed at our center using the standard procedure (no device for guide wire positioning).
  This control group should have registered al parameters and variables to be studied.
  Interventions: Procedure: Scaphoid fixation using standard procedure
- Case Patients: Prospective series of ten patients on which the external 3D guide system will be used.
  Interventions: Device: Scaphoid fixation using 3D device

INTERVENTIONS:
Device: Scaphoid fixation using 3D device — A headless screw inserted percutaneously from the volar aspect of the scaphoid in a retrograde manner using a customised 3D exoesqueleton guide
  Groups: Case Patients
Procedure: Scaphoid fixation using standard procedure — A headless screw inserted percutaneously from the volar aspect of the scaphoid in a retrograde manner without using the 3D device (standard procedure)
  Groups: Control Patients

SUMMARY:
The investigators want to analyse the advantages of using a 3D constructed prototype from a previous CT Scan to model an external customised guide por percutaneous Scaphoid fixation.

The investigators hypothesise that the usage of this device will shorten surgery time, radiation for the surgery team and optimise the percutaneous screw trajectory inside of the scaphoid bone.

DETAILED DESCRIPTION:
To carry out this analysis the investigators will recruit 10 patients who present with an acute fracture of the Scaphoid bone type B1 and B2 (Herbert Classification).

A CT Scan will be performed and a 3D exoesqueleton model printed, previously deciding the position of the fixation screw inside of the bone and adding a cannulated sleeve in the volar aspect of the exoesqueleton to insert the initial positional guide wire for surgery.

Surgery time, surgery radiation exposure and screw positioning will be recorded and compared to 10 control patients operated following standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* Acute scaphoid fracture (Herbert B1 B2)

Exclusion Criteria:

* Concomitant fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an Scaphoid acute fracture that requires surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-03-25 (Actual); Primary Completion 2019-03-25 (Estimated); Study Completion 2019-03-29 (Estimated)

PRIMARY OUTCOMES:
Screw Position | 1st day Xray
  Correct position of screw inside of the scaphoid

SECONDARY OUTCOMES:
Surgery time | 1st day
  time from beginning to completion of surgery
xray exposure | 1st day
  radiation exposure during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francesc A Marcano Fernandez, MD, Principal Investigator — Hospital parc tauli Sabadell
Locations (1):
- Corporación sanitaria Parc Taulí de Sabadell, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No